CLINICAL TRIAL: NCT03204565
Title: Effectiveness of Adjunctive Hyaluronic Acid Application in Coronally Advanced Flap in Miller Class I Single Gingival Recession Sites
Brief Title: Effectiveness of Adjunctive Hyaluronic Acid Application in Coronally Advanced Flap in Single Gingival Recession Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Chairman Section of Periodontics Director of Master Program in Periodontics, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #2538/15
Record Dates: First submitted 2017-06-25; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Gingival Recession
Keywords: gingival recession, clinical trial(s).
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- CAF + HA (Test) (Experimental): coronally advanced flap with hyaluronic acid
  Interventions: Procedure: coronally advanced flap; Device: hyaluronic acid
- CAF (control) (Active Comparator): coronally advanced flap alone
  Interventions: Procedure: coronally advanced flap

INTERVENTIONS:
Procedure: coronally advanced flap — coronally advanced flap alone (CAF- control)
Device: hyaluronic acid — hyaluronic acid associated to coronally advanced flap (CAF + HA- test)
  Arms: CAF + HA (Test)

SUMMARY:
The purpose of this randomized controlled clinical trial (RCT) is to determine the efficacy hyaluronic acid (HA) in combination with the coronally advanced flap (CAF) for the treatment of single gingival recession site.

The hypothesis is that HA will result in improved the clinical outcomes and will reduce the pos-operative morbidity

DETAILED DESCRIPTION:
Gingival recession is a common clinical finding in patients with high standards of oral hygiene and can be found in more than 90% of patients. Buccal exposure of roots with aesthetic impairments and dentinal hypersensitivity The ultimate goal of root coverage procedures is the complete coverage of the recession defect with an aesthetic appearance comparable to adjacent healthy soft tissues in combination with physiological probing pocket depths.Several surgical techniques have already provided good results and have been shown to attain root coverage at individual recession sites these different methods.To date, connective tissue grafts (CTG) and enamel matrix derivatives (EMD) in conjunction with a coronally advanced flap (CAF) have been shown to provide the highest probability of obtaining complete root coverage (CRC) in Miller class I and II single gingival recession as compared to CAF alone.

Hyaluronic acid (HA) is a major component of the extracellular matrix in almost all tissues. The primary role of HA is to bind water and to permit the transportation of key metabolites and therefore to maintain the structural and homeostatic integrity of these tissues.

In vitro and animal studies have demonstrated that hyaluronic acid have many properties that are essential for tissue regeneration and wound healing.

However, to the best of our knowledge, there have been limited clinical application studies in the field of root coverage procedures performed and still no consistent published data with longer follow-ups on the usage of HA are available.

Therefore, the aim of this randomized controlled clinical trial (RCT) was to evaluate the potential benefit of the adjunctive use of HA in combination with a coronally advanced flap (CAF) and to compare the outcomes with CAF alone, when treating single Miller Class I gingival recessions.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) < 15% (measured at four sites per tooth)
* presence of at least one buccal recession (depth ≥2 mm) classified as Miller Class I. Only gingival recession sites localized in the anterior area of the maxillary or mandibular arch (central and lateral incisors, canine and first and second premolars) and associated with aesthetic problems and/or dental hypersensitivity were enclosed
* gingival recession with at least 1 mm of keratinized tissue (KT) apical to the recession
* presence of a clearly identifiable cemento-enamel junction (CEJ), 10) no teeth with prosthetic crown or restoration with the cervical edge in the CEJ area

Exclusion Criteria:

* systemic diseases or pregnancy
* smokers
* systemic antibiotic therapy in the last 6 months
* active periodontal disease with a sites (probing pocket depth <4 mm and no bleeding on probing)
* history of mucogingival or periodontal surgery at the experimental site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Recession reduction (RecRed) | baseline and 18 months
  Changes in recession depth between initial and final. Measured in mm

SECONDARY OUTCOMES:
Post-operative morbidity (pain, swelling and discomfort) | 7 days
  With an evaluation questionnaire. The interviewer assessed patient's pain, swelling and discomfort at 7 days after procedure using visual analogue scale (VAS) ranging from 0 (no pain/swelling/discomfort) to 10 (maximal pain/swelling/discomfort).
Complete root coverage (CRC) | 18 months
  Assessed as percentage of sites with complete root coverage
Mean root coverage (MRC) | 18 months
  Assessed as percentage of mean root coverage for each group.
Probing pocket depth (PPD) | baseline and 18 months
  Changes in PPD between initial and final. Measured in mm
Clinical attachment level gain (CAL-Gain) | baseline and 18 months
  Difference between CAL initial and final. Measured in mm
Width of keratinized tissue (KT) | baseline and 18 months
  Changes in KT between initial and final. Measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD,DDS,MS, Study Director — University La Sapienza, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moseley R, Waddington RJ, Embery G. Hyaluronan and its potential role in periodontal healing. Dent Update. 2002 Apr;29(3):144-8. doi: 10.12968/denu.2002.29.3.144. PMID 11989392
- [Background] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000
- [Background] Pilloni A, Paolantonio M, Camargo PM. Root coverage with a coronally positioned flap used in combination with enamel matrix derivative: 18-month clinical evaluation. J Periodontol. 2006 Dec;77(12):2031-9. doi: 10.1902/jop.2006.050390. PMID 17209788
- [Background] Tatakis DN, Chambrone L, Allen EP, Langer B, McGuire MK, Richardson CR, Zabalegui I, Zadeh HH. Periodontal soft tissue root coverage procedures: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S52-5. doi: 10.1902/jop.2015.140376. Epub 2014 Oct 15. PMID 25315018
- [Background] Kumar R, Srinivas M, Pai J, Suragimath G, Prasad K, Polepalle T. Efficacy of hyaluronic acid (hyaluronan) in root coverage procedures as an adjunct to coronally advanced flap in Millers Class I recession: A clinical study. J Indian Soc Periodontol. 2014 Nov-Dec;18(6):746-50. doi: 10.4103/0972-124X.147411. PMID 25624632
- [Background] Ferguson EL, Roberts JL, Moseley R, Griffiths PC, Thomas DW. Evaluation of the physical and biological properties of hyaluronan and hyaluronan fragments. Int J Pharm. 2011 Nov 25;420(1):84-92. doi: 10.1016/j.ijpharm.2011.08.031. Epub 2011 Aug 22. PMID 21884772
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] Weigel PH, Frost SJ, McGary CT, LeBoeuf RD. The role of hyaluronic acid in inflammation and wound healing. Int J Tissue React. 1988;10(6):355-65. PMID 2855633